CLINICAL TRIAL: NCT01258049
Title: A Phase III, Randomised, Open Labelled, Active Controlled, Multi Centre, Superiority Trial of ArTiMist™ Versus Intravenous Quinine in Children With Severe or Complicated Falciparum Malaria, or Uncomplicated Falciparum Malaria With Gastrointestinal Complications.
Brief Title: Superiority of ArTiMist Versus Quinine in Children With Severe Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Proto Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART004
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Plasmodium infections; Remittent fever; Artemether; Artemesinins; Quinine; Malaria; Protozoan infections; sublingual drug delivery; Parasitic disease; Antiprotozoan agents
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Protozoan Infections; Parasitic Diseases | interventions — Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ArTiMist (Experimental)
  Interventions: Drug: Artemether Sublingual Spray
- Quinine (Active Comparator)
  Interventions: Drug: Quinine

INTERVENTIONS:
Drug: Artemether Sublingual Spray — Artemether sublingual spray administered at 3 mg/kg (milligrams per kilogram) at specified timepoints
  Other Names: ArTiMist
  Arms: ArTiMist
Drug: Quinine — Quinine administered intravenously, 20 mg/kg loading dose followed by 10 mg/kg every eight hours
  Arms: Quinine

SUMMARY:
The purpose of this study is to demonstrate that ArTiMist (sublingual artemether spray) is better than intravenous quinine in reducing parasite counts by >= 90% within 24 hours after the start of treatment in children with severe malaria, or uncomplicated malaria with gastrointestinal complications

DETAILED DESCRIPTION:
Malaria causes significant morbidity and mortality in children in developing countries, despite the availability of highly effective antimalarial therapy. One of the key contributing factors is the delay in the initiation of treatment.

ArTiMist is a sublingual formulation of the established antimalarial treatment, artemether. In previous studies good bioavailability has been demonstrated. In an exploratory study (ART003) ArTiMist demonstrated a non statistically significant improvement of 26% (when compared to intravenous quinine) in the numbers of patients experiencing a parasite reduction of >= 90% within 24 hours of the initiation of treatment.

This Phase 3 study is being conducted to establish whether treatment with ArTiMist in children with severe falciparum malaria or uncomplicated falciparum malaria with gastrointestinal complications is at least 20% superior in providing parasitological success (defined as >= 90% reduction in parasite count at 24 hours after start of treatment) when compared to intravenous quinine.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's legally acceptable representative has provided informed consent and the patient has assented (where relevant) to participation in the trial
2. The patient is a child that weighs between 5.00 kg and 15.00 kg inclusive
3. The patient has falciparum malaria as evidenced by thick or thin blood smears of ≥ 500 P Falciparum per mcl (patients with mixed infections may be included provided ≥ 500 P Falciparum per mcl)
4. The patient has either:

   * severe or complicated falciparum malaria as determined by the investigator based on the WHO criteria for severity, and/or
   * uncomplicated falciparum malaria but is unable to tolerate oral medication as a result of gastrointestinal complications such as vomiting or diarrhoea.

Exclusion Criteria:

1. The patient's legally acceptable representative does not provide informed consent for participation, or the child if capable, does not assent to participation in the trial.
2. Ability to tolerate oral therapy
3. Patient has received any antimalarial therapy within the 7 days prior to first study drug administration.
4. Patient has evidence of significant co-infections (this does not include mixed Plasmodium infections).
5. Patient has a contraindication, allergy or is otherwise intolerant to either artemether or quinine .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl Bendel, MBChB MFPM, Study Chair — Xidea Solutions Limited
Locations (3):
- Centre National de Recherche et de Formation sur le Paludisme (CNRFP), Ouagadougou, Burkina Faso
- Navrongo Health Research Centre, Navrongo, Navrongo, Ghana
- Rwinkwavu District Hospital, Rwinkwavu, Eastern Province, Rwanda

REFERENCES:
- [Derived] Bendel D, Rulisa S, Ansah P, Sirima S. Efficacy of a novel sublingual spray formulation of artemether in African children with Plasmodium falciparum malaria. Antimicrob Agents Chemother. 2015 Nov;59(11):6930-8. doi: 10.1128/AAC.00243-15. Epub 2015 Aug 24. PMID 26303805

RESULTS

PARTICIPANT FLOW:
Groups:
- ArTiMist: Doses of 3 mg/kg were administered sublingually at: 0 h, 8 h, 24 h, 36 h, 48 h, and 60 h. Following the initial six doses, subjects could, at the discretion of the Investigator receive a further four daily doses of 3 mg/kg ArTiMist™ to complete a seven day treatment course, or be converted to another suitable treatment or a suitable course of combination therapy in accordance with national drugs policy where applicable.
- Quinine: A loading dose of 20 mg/kg was given over four hours and thereafter 10 mg/kg was given every eight hours until the subject was able to swallow. Thereafter, patients were given quinine syrup or crushed tablets (10 mg/kg every eight hours) or another suitable treatment to ensure they received at least seven days of therapy, or be converted to another suitable treatment or a suitable course of combination therapy, in accordance with national drugs policy where applicable.
Period: Overall Study
Arm/Group | ArTiMist | Quinine
Started | 77 | 74
Completed | 75 | 72
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ArTiMist | Quinine | Total
Number analyzed (Participants) | 77 | 74 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.8 (1.34) | 2.5 (1.23) | 2.6 (1.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 79
  Male | 37 | 35 | 72
Region of Enrollment [Number; unit: participants]
  Ghana | 25 | 25 | 50
  Burkina Faso | 25 | 25 | 50
  Rwanda | 27 | 24 | 51
Disease Definition - Severe or complicated malaria [Number; unit: participants]
  Severe or complicated malaria | 49 | 51 | 100
  Uncomplicated malaria with GI complications | 28 | 23 | 51
Weight [Mean (Standard Deviation); unit: kg] | 11.7 (2.4) | 11.2 (2.5) | 11.4 (2.5)
Pulse rate [Mean (Standard Deviation); unit: bpm] | 146 (20.2) | 147 (26.3) | 146 (23.3)
Tympanic Temperature [Mean (Standard Deviation); unit: Degrees Centigrade] | 38.6 (1.1) | 38.6 (1.0) | 38.6 (1.1)
Respiratory Rate [Mean (Standard Deviation); unit: breaths/min] | 36.7 (11.0) | 35.9 (11.3) | 36.3 (11.2)
Blantyre Coma Scale [Number; unit: participants] — Blantyre Coma scale scores out of 5, full consciousness, by adding the scores of the following 3 domains. Any score ≤ 4 is considered abnormal,
  Eye Movement
  1 Watches or follows 0 Fails to watch or follow
  Best Motor Response 2 Localizes painful stimulus 1 Withdraws limb from painful stimulus 0 No response or inappropriate response
  Best Verbal Response 2 Cries appropriately with pain, or if verbal, speaks
  1 Moan or abnormal cry with pain 0 No vocal response with pain
  participants
    5 | 60 | 53 | 113
    < 5 | 17 | 21 | 38
Parasite Counts [Mean (Standard Deviation); unit: p falciparum /mcl] | 133884 (129715) | 155321 (202213) | 144602 (165964)
Parasite Count (median) [Median (Full Range); unit: p falciparum /mcl] | 86572 [279 to 515556] | 66077 [1225 to 843746] | 76325 [279 to 843746]

OUTCOME MEASURES:

1. Primary Outcome: Parasitological Success (MITT)
Description: Parasitological success defined as a reduction in parasite count of ≥ 90% of baseline at 24 hours after the first dose
Time Frame: 24 hours after start of treatment
Population: The Modified Intention to Treat (MITT) population included all randomised subjects who received at least one dose of study medication and had evaluable parasite counts at 24 hours after first dosing.
  7 subjects for ArTiMist and 3 subjects for quinine were excluded due to no baseline or 24 h parasite count
Measure: Number; unit: participants
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
participants
  Success | 66 | 28
  Not Success | 4 | 43
Statistical Analysis 1: Comparison: ArTiMist vs Quinine; In ART003, the parasite success rate for quinine was 67.7%. On the assumption that the parasite success rate was 70% for quinine in this study and in order to demonstrate that ArTiMist™ is superior to quinine by at least 20% the success rate for ArTiMist™ should be at least 90%. Using these figures, and assuming a power of 80%, an alpha of 0.05 (two sided) and based on an equal allocation to the ArTiMist™ and quinine treatment arms, the number of subjects (n) required on each treatment was 59; Test type: Superiority or Other; p < 0.005, Regression, Logistic; Percentage Difference = 54.85, 95% CI 2-sided [42.25 to 67.45]

2. Secondary Outcome: Parasite Clearance Time (PCT) [MITT Population]
Description: Parasite clearance time (PCT). Time in hours from the initiation of therapy until the first of two successive parasite negative smears (zero parasite counts) are obtained
Time Frame: 28 days after start of treatment
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
hours | 30.29 (13.21) | 68.30 (98.04)
Statistical Analysis 1: Comparison: ArTiMist; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Final Values) = -38.97, 95% CI 2-sided [-62.22 to -15.72]

3. Secondary Outcome: PCT 90 [MITT Population]
Description: Time for parasite counts to fall by 90%
Time Frame: 28 days after start of treatment
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
hours | 15.02 (5.82) | 27.93 (18.03)
Statistical Analysis 1: Comparison: ArTiMist vs Quinine; Test type: Superiority or Other; p < 0.005, ANCOVA; Mean Difference (Final Values) = -12.91, 95% CI 2-sided [-17.38 to -8.44]

4. Secondary Outcome: PCT 50 [MITT Population]
Description: Time for parasite counts to fall by 50%
Time Frame: 28 days after start of treatment
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
hours | 9.42 (5.72) | 18.58 (9.19)
Statistical Analysis 1: Comparison: ArTiMist vs Quinine; Test type: Superiority or Other; p < 0.005, Regression, Cox; Mean Difference (Final Values) = -9.16, 95% CI 2-sided [-11.71 to - 6.61]

5. Secondary Outcome: PRR 24 [MITT Population]
Description: The percentage reduction in parasite counts 24 hours after first dose
Time Frame: 28 days after start of treatment
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
percentage of baseline | 98.2 (6.12) | 44.5 (114.27)
Statistical Analysis 1: Comparison: ArTiMist vs Quinine; Test type: Superiority or Other; p < 0.005, ANCOVA; Mean Difference (Final Values) = 54.02, 95% CI 2-sided [27.05 to 80.98]

6. Secondary Outcome: PRR 12 [MITT Population]
Description: The percentage reduction in parasite counts 12 hours after first dose
Time Frame: 28 days after start of treatment
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
percentage of baseline | 47.6 (70.28) | -132.2 (765.92)
Statistical Analysis 1: Comparison: ArTiMist vs Quinine; Test type: Superiority or Other; p = 0.06, ANCOVA; Mean Difference (Final Values) = 174.09, 95% CI 2-sided [-10.44 to 358.61] — mean parasite counts increased in the first 12 hours for patients on quinine treatment

7. Secondary Outcome: Fever Clearance Time (FCT)
Description: Time in hours from the initiation of therapy until the disappearance of fever (tympanic temperature < 38.0) that lasted at least 24 hours.
Time Frame: 28 days after start of treatment
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
hours | 42.6 (34.47) | 41.6 (22.73)
Statistical Analysis 1: Comparison: ArTiMist vs Quinine; Test type: Superiority or Other; p = 0.86, Regression, Cox; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-10.16 to 12.08]

8. Secondary Outcome: Complete Cure Rate
Description: The complete resolution of clinical signs and symptoms, malaria-related laboratory abnormalities, and elimination of asexual parasites by Day 7, with no recurrence up to Day 28 (+/- 2 days), and the 48h parasite count to be < 25% of baseline with no clinical deterioration
Time Frame: 28 days after the start of treatment
Population: For some subjects, this endpoint was not evaluable and/or not all data was received.
Measure: Number; unit: participants
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 55 | 63
participants
  Cure | 41 | 46
  No Cure | 14 | 17
Statistical Analysis 1: Comparison: ArTiMist vs Quinine; Test type: Superiority or Other; p = 0.99, Regression, Logistic; Percentage Difference = 0.99, 95% CI 2-sided [0.42 to 2.36]

9. Secondary Outcome: Early Treatment Failure
Description: Early treatment failure is indicated by one or more of the following:
  * Parasite count on Day 2 > Day 0, irrespective of temperature
  * Parasite count on Day 3 > 0 with tympanic temperature ≥ 38.0°C
  * Parasite count on Day 3 ≥ 25% of baseline
  * Administration of rescue antimalarial treatment
Time Frame: Three days after the start of treatment
Measure: Number; unit: participants
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
participants | 0 | 14

10. Secondary Outcome: Late Clinical Failure
Description: * Signs of severe malaria on any day between Day 4 and Day 28 in the presence of parasitaemia, without previously meeting any of the criteria of early treatment failure
  * Presence of parasitaemia and tympanic temperature ≥ 38.0°C (or history of fever), on any day between Day 4 and Day 28, without previously meeting any of the criteria of early treatment failure
Time Frame: 28 days after the start of treatment
Measure: Number; unit: participants
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
participants | 3 | 1

11. Primary Outcome: Parasitological Success (PP)
Description: Parasitological success defined as a reduction in parasite count of ≥ 90% of baseline at 24 hours after the first dose
Time Frame: 24 hours after start of treatment
Population: The Per Protocol (PP) population included the subjects in the MITT population who had received at least 80% of doses up to the time of discharge from the hospital, had evaluable data up to and including Day 28 and had no major protocol violations.
Measure: Number; unit: participants
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 68 | 69
participants
  Success | 65 | 28
  Not Success | 3 | 41
Statistical Analysis 1: Comparison: ArTiMist vs Quinine; Test type: Superiority or Other; p < 0.005, Regression, Linear; Percentage Difference = 55.01, 95% CI 2-sided [42.44 to 67.58]

12. Secondary Outcome: Late Parasitological Failure
Description: o Parasitaemia on any day from Day 7 to Day 28 and tympanic temperature ≤ 38.0°C
Time Frame: 28 days after the start of treatment
Measure: Number; unit: participants
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
participants | 12 | 14

13. Secondary Outcome: Time to Return to Full Consciousness
Description: Time in hours to return to full consciousness (Blantyre Coma Scale = 5), if level of consciousness is reduced (Blantyre Coma Scale <5) prior to dosing or within 24hours of first dosing.
  For the Blantyre Coma Scale
  Total - maximum 5, eye movement - maximum 1, best motor response - maximum 2, best verbal response - maximum 2
Time Frame: 28 days after start of treatment
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
hours | 20.8 (9.58) | 23.0 (16.52)

14. Secondary Outcome: Time to Return to Normal Per os Status
Description: Time in hours to return to normal per os status. Normal per os was when the investigator considered the patient to be able to eat and drink normally.
Time Frame: 28 days after start of treatment
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
hours | 22.1 (12.89) | 25.3 (16.28)

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events, of Possible, Probably and Definite Causalities
Time Frame: 28 days after start of treatment
Measure: Number; unit: participants
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
participants | 5 | 6

16. Secondary Outcome: Number of Deaths or Neurological Sequelae at Day 28
Time Frame: 28 days after start of treatment
Measure: Number; unit: participants
Arm/Group | ArTiMist | Quinine
Number analyzed (Participants) | 70 | 71
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of signing informed consent until the final study visit. Adverse events that started or worsened after start of treatment were considered Treatment Emergent.
Arm/Group | ArTiMist | Quinine
Serious Adverse Events (participants affected / at risk) | 4/77 | 10/74
Other Adverse Events (participants affected / at risk) | 43/77 | 44/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ArTiMist (N=77) | Quinine (N=74)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 7 (7)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cerebral Malaria (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ArTiMist (N=77) | Quinine (N=74)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 12 (12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
Pyrexia (General disorders) | 7 (7) | 6 (6)
Malaria (Infections and infestations) | 17 (17) | 14 (14)
Respiratory Tract Infection (Infections and infestations) | 7 (7) | 3 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No